CLINICAL TRIAL: NCT02031562
Title: Geriatric Balance and Low Back Pain and Balance Assessment and Management
Brief Title: Geriatrics Balance and Low Back Pain Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Collaborators: St. Louis University (Other)
Responsible Party: Principal Investigator, Dennis Enix, DC, MBA, Associate Professor, Logan College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD1002090203; R18HP15125 (Other Grant/Funding Number: HRSA)
Record Dates: First submitted 2013-12-18; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Distorted Balance; Low Back Pain
Keywords: Balance; Falls; Low back pain; Geriatric
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Chiropractic; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chiropractic (Active Comparator): Chiropractic
  Interventions: Other: chiropractic
- Physical therapy (Active Comparator): Physical therapy
  Interventions: Other: physical therapy

INTERVENTIONS:
Other: chiropractic — chiropractic
  Arms: Chiropractic
Other: physical therapy — physical therapy
  Arms: Physical therapy

SUMMARY:
This study evaluates the effect of standard of care treatments (physical therapy versus manual therapy) in older adult patients who have balance problems with or without low back pain.

DETAILED DESCRIPTION:
This study uses a randomized controlled research design and will enroll up to three hundred patients. Treatment will take place in outpatient facilities. It is hypothesized that among older adults with low back pain manual therapy will reduce low back pain and improve balance more than physical therapy; and that among older adults without low back pain manual therapy and physical therapy will be equally efficacious in improving balance. The results of this study will help to further define effective treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 60-85
* self reported balance problems
* With or with out low back pain.

Exclusion Criteria:

* History of recent fracture or surgery of lumbar spine, pelvis, hip or femur
* History of recent neoplasm (minor skin cancers are not excluded)
* Acute infectious disease
* Chronic low back pain persisting for >8 weeks
* Severe disabling health problems so that patient is not ambulatory
* Non-mechanical low back pain
* Recent unstable peripheral vascular disease and or cardiac disease requiring recent hospitalization < 6 months ago
* Patients with balance problems related to the following: Meniere's disease, vertigo, or vestibular disorders
* Recent history of self reported substance abuse
* Ongoing treatment for balance problems or low back pain by chiropractor, physical therapist, or orthopedic physician or other physician.
* Current use of medication from the following categories: antipsychotics, anxiolytics, and sedative/hypnotics

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2009-10; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in patient balance parameters at baseline, 6 weeks and 12 weeks. | Baseline, week 6 and week 12.
  Participants complete functional performance tests and self-report questionnaires related to balance, pain, and quality of life. Testing is performed at baseline, after 6 weeks of care, and at 12 weeks. Balance tests included the Berg Balance Scale, The Timed Get up and Go (TGUG) test, Performance-oriented mobility assessment (POMA), NeuroCom Balance assessment tests which included the Limits of Stability (LOS) Test and Modified Clinical test for the sensory integration of Balance (Mod CTSIB).

SECONDARY OUTCOMES:
Change in patient pain levels at baseline, 6 weeks and 12 weeks. | Baseline, week 6 and week 12.
  Self reported questionnaires include the Falls Efficacy Scale (FES), Tampa Kinesiophobia Scale, Visual analogue scale (VAS), the 21-point Box Pain Scale, the Oswestry Questionnaire, SF-36 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dennis E Enix, DC, MBA, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States